CLINICAL TRIAL: NCT06382376
Title: Four-quadrant Transversus Abdominis Plane Block Versus Intrathecal Morphine in Gynecological Cancer Surgeries: a Single-center Retrospective Study.
Brief Title: The Effect of Analgesia Methods Applied in Gynecological Cancer Surgeries on Postoperative Analgesia
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Duygu Akyol, Principal Investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: 2024-60
Record Dates: First submitted 2024-04-20; First posted 2024-04-24 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Gynecological Cancer Surgery; Regional Anesthesia Morbidity
Keywords: gynecological cancer surgery; periferal block; neuraxial block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Intrathecal morphine administered group: Group 1: Intrathecal morphine administered group
  Interventions: Procedure: Intrathecal morphine administered group, Four quadrant transversus abdominis plane block applied group
- Group 2: Four quadrant transversus abdominis plane block applied group: Group 2: Four quadrant transversus abdominis plane block applied group
  Interventions: Procedure: Intrathecal morphine administered group, Four quadrant transversus abdominis plane block applied group

INTERVENTIONS:
Procedure: Intrathecal morphine administered group, Four quadrant transversus abdominis plane block applied group — Intrathecal morphine administered group and Four quadrant transversus abdominis plane block applied group
  Other Names: Group 1: Intrathecal morphine administered group; Group 2: Four quadrant transversus abdominis plane block applied group

SUMMARY:
The aim of this study is to compare the effectiveness of intrathecal morphine and four-quadrant transversus abdominis plane block applied for postoperative analgesia in gynecological cancer surgeries.

The key question(s) it aims to answer are:

[Is intrathecal morphine more effective in postoperative analgesia?] Patients who underwent gynecological cancer surgery were examined retrospectively. The investigators evaluated the effect of intrathecal morphine and four-quadrant transversus abdominis plane block applied for postoperative analgesia on pain scores and postoperative opioid use.

DETAILED DESCRIPTION:
Our study was designed retrospectively. The investigators evaluated analgesia methods in patients who underwent laparoscopic or open surgery due to gynecological cancer between June 2023 and December 2023. The investigators evaluated the effect of intrathecal morphine and four-quadrant transversus abdominis plane block on postoperative analgesia and opioid use.

Group 1: Intrathecal morphine administered group Group 2: Four quadrant transversus abdominis plane block applied group

ELIGIBILITY:
Inclusion Criteria:

* 18 years

  * Patients who have undergone gynecological cancer surgery

Exclusion Criteria:

* <18 years
* Those with missing data

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Between June 1, 2023 and December 1, 2023, 71 patients over the age of 18 who underwent surgery for ASA II and III gynecological cancer, to whom we applied intrathecal morphine or four-quadrant transversus abdominis plane block (TAPB) from peripheral nerve blocks for postoperative analgesia, were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
postoperative numerical rating scale | 24 hours postoperatively
  Our primary aim was to evaluate numerical rating scale at 24 hours postoperatively. numerical rating scale(NRS) was used to assess postoperative pain. NRS values were recorded For example, 0-10 where 0 is no pain and 10 is the worst pain imaginable.

SECONDARY OUTCOMES:
postoperative opioid use | 24 hours postoperatively
  Our secondary aim was to evaluate opioid demand and consumption amounts in the postoperative 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Akyol, Principal Investigator — Başakşehir Çam & Sakura City Hospital
Locations (1):
- Başakşehir Çam and Sakura City Hospital, Istanbul, Basaksehir, Turkey (Türkiye)

REFERENCES:
- [Result] Black KA, Nelson G, Goucher N, Foley J, Pin S, Chong M, Ghosh S, Bisch SP. Effect of transversus abdominis plane block on postoperative outcomes in gynecologic oncology patients managed on an Enhanced Recovery After Surgery pathway. Gynecol Oncol. 2023 Nov;178:1-7. doi: 10.1016/j.ygyno.2023.09.003. Epub 2023 Sep 18. PMID 37729808
- [Result] Niraj G, Kelkar A, Hart E, Kaushik V, Fleet D, Jameson J. Four quadrant transversus abdominis plane block and continuous transversus abdominis plane analgesia: a 3-year prospective audit in 124 patients. J Clin Anesth. 2015 Nov;27(7):579-84. doi: 10.1016/j.jclinane.2015.07.005. Epub 2015 Aug 28. PMID 26319886
- [Result] Pirie K, Traer E, Finniss D, Myles PS, Riedel B. Current approaches to acute postoperative pain management after major abdominal surgery: a narrative review and future directions. Br J Anaesth. 2022 Sep;129(3):378-393. doi: 10.1016/j.bja.2022.05.029. Epub 2022 Jul 6. PMID 35803751
- [Result] Meylan N, Elia N, Lysakowski C, Tramer MR. Benefit and risk of intrathecal morphine without local anaesthetic in patients undergoing major surgery: meta-analysis of randomized trials. Br J Anaesth. 2009 Feb;102(2):156-67. doi: 10.1093/bja/aen368. PMID 19151046